# **Cover Page for Protocol**

| Sponsor-Investigator: | Diana Jalal |
|-----------------------|--------------------------------------|
| NCT Number: | NCT03597568 |
| Unique Protocol ID: | 201806073 |
| Official Title: | Effect of resveratrol on endothelial |
| | function in patients with CKD and |
| | diabetes: A randomized controlled |
| | trial |
| Document Date: | 23 February 2024 |

# **Background and significance**

Patients with chronic kidney disease (CKD) have an exceptionally high risk for cardiovascular disease (CVD) and are 10 times more likely to die from CVD prior to requiring dialysis or kidney transplantation (1). Multiple studies have shown CKD to be an independent risk factor for cardiovascular events and mortality (2-6). Diabetes mellitus is the most common cause of CKD and is believed to contribute to a significant portion of the CVD with CKD (7). Indeed, patients with CKD and diabetes have a disproportionally higher risk for CVD when compared with patients with diabetes who do not have CKD (8). Thus, it is paramount that we explore therapies that may ultimately reduce the burden of CVD in

those with CKD and diabetes.

Endothelial dysfunction via brachial artery flow mediated dilation (BA-FMD), is a reliable and non-invasive vascular assessment, which has been shown to predict CVD prospectively in a wide variety of 'at-risk' and diseased populations, including individuals with CKD (9). Preliminary data by our group demonstrates that endothelial function via BA-FMD test is significantly lower in individuals with CKD and diabetes as compared to those with CKD but without DM (**Fig** 1). These findings suggest that the etiology of DM within CKD patients appears to exacerbate the condition more so than CKD alone.

Experimental studies, suggest that resveratrol (a widely-available nutraceutical) inhibits inflammation and restores endothelial nitric oxide (NO) *in vitro* (9-11) and *in vivo* (12,13).



In this pilot study, we will evaluate if resveratrol supplementation improves endothelial function and oxidative stress in those with CKD and diabetes.

## Study Design

25 subjects with stage 3 CKD and diabetes will randomized to receive either resveratrol first then matching placebo or placebo first then resveratrol in a randomized cross over study. Resveratrol will be prescribed at 400 mg per day. The treatment resveratrol or placebo will be for 6 weeks and separated by a 2 week washout period.

The inclusion criteria are shown in **Table 1**.

| Table 1 | |
|---|---|
| Inclusion Criteria | Exclusion Criteria |
| Age 45-80 years old | Consuming >2 glasses/day red wine and/or taking resveratrol or vitamin C supplement in the past 12 months |
| CKD stage 3 (CKD-EPI eGFR:<br>30-60 mL/min/1.73m²) on 2<br>occasions ≥3 months apart | Life expectancy <1 year |
| Type II DM | Pregnant, breastfeeding, or unwilling to use adequate birth control |
| angiotensin converting enzyme inhibitor or angiotensin II receptor blocker for ≥3 months prior to the study | Uncontrolled hypertension; blood pressure >140/90 |
| Able to give informed consent | Severe liver disease |
| | Severe congestive heart failure |
| | Hospitalization within the last 3 months |
| | Active infection or antibiotic therapy |
| | Immunosuppressive therapy within the last year |
| | Uncontrolled DM with A1C > 8.5 |
| | Currently taking anticoagulants including the following: coumadin, dalteparin, enoxaparin, heparin, and plavix. |
| | Severe systolic heart failure |
| | Currently partaking in another research study |

Our rational for RSV dose is that: 1) it is available commercially at 400 mg and 2) recent studies utilizing RSV suggest that this dose is safe and does not result in serious side effects (14, 15).

The study is registered with clinicaltrials.gov

Institutional Review Board was obtained. The informed consent will detail the risks associated with the study drug and with all the study procedures.

## Detailed study sessions

All study procedures will be conducted at UIHC Clinical Research Unit (CRU) and all experimental testing measurements will be conducted after an overnight fast as well as refraining from exercise and caffeine prior to testing.

**Session 1:** Informed consent and screening questionnaire for inclusion and exclusion criteria including confirmation of stage 3 CKD on 2 separate occasions in the last 6 months. All women in child-bearing age will undergo pregnancy test at this visit. In addition, all participants will complete a 7-day physical activity recall.

#### Session 2:

- Blood pressure at rest
- · Endothelial cell sampling
- · Blood sampling for fasting lipid profile
- Blood sampling for hemoglobin A1C
- · Blood sampling for levels of RSV and its metabolites
- Blood sampling for basic metabolic profile and estimated GFR including cystatin C
- Blood sampling for circulating markers of inflammation and oxidative stress (oxLDL)
- Urine sampling (random) for albumin/creatinine ratio (ACR)
- Evaluation of EDD and EID by measurements of BA-FMD and nitroglycerin-mediated dilation (NMD)
- Start study drug after this visit

**Session 3:** will include the same measurements as Session 2. In addition, it will include the following:

- Physical activity questionnaire
- Pill count
- Safety monitoring:
  - Completion of an adverse event questionnaire
  - Update medication list

**Sessions 4 and 5:** will involve the exact same procedures as Sessions 2 & 3 above except it will involve the other study drug being ingested for 6 weeks (resveratrol or placebo).

### Outcome measurements

1. Measurements of endothelial dependent and independent dilation: Endothelial dependent dilation (EDD) of the brachial artery (BA-FMD) will be measured at the Cardiovascular Research Lab in the Clinical Research Unit (CRU) at the University of Iowa by principal investigator using high-resolution Doppler ultrasonography as described originally by Celermajer et al (16,17). Electrocardiogram (ECG) gated end-diastolic ultrasound images and Doppler flow of the artery will be acquired during baseline and FMD and conditions. Briefly, and after 15 minutes of quiet supine rest, the vascular reactivity of the brachial artery will be assessed as based on the following: 1) two minutes of baseline hemodynamics followed by inflation of a rapidly inflating pneumatic pediatric cuff wrapped around the maximal circumference of the forearm to a pressure of 240 mmHg for 5 min, and 2) rapid deflation of the cuff after five minutes. A commercially available software package will be used to acquire and analyze ECG-gated brachial artery diameters. Endothelial independent dilation (EID) will also be determined by measuring brachial artery dilation for 10 minutes after administration of sublingual nitroglycerin (0.4 mg). BA-FMD

(pre- vs. post-intervention) will be calculated as the % change from baseline and compared against the placebo condition.

- 2. <u>Systemic markers of oxidative stress</u>: oxidized low density lipoprotein (LDL) cholesterol (ALPCO Diagnostics, Catalog #30-7810) will be quantified using commercially available enzyme-linked immunosorbent assays performed according to kit instructions.
- 3. Endothelial cell sampling and cell protein expression: This technique will be done by a trained/qualified individual at the UI CRU. Briefly, J-wires will be advanced into an antecubital vein and withdrawn. Cells will be recovered by standard techniques (18). Collected cells will be fixed with 3.7% formaldehyde and plated on slides. After blocking nonspecific binding sites with 5% donkey serum, cells are incubated with the primary antibody and with CY3-conjugated secondary antibodies. Slides will be systematically scanned to identify endothelial cells (positive VE-Cadherin) and nuclear integrity confirmed using 4',6'-diamidino-2-phenylindole hydrochloride staining. Once endothelial cells with intact nuclei are identified, images will be captured and then analyzed to quantify the intensity of CY3 staining (i.e., average pixel intensity). Values for each sample will be reported as ratios of endothelial cell protein expression/human umbilical vein endothelial cell (HUVEC) to account for any variation in the staining procedure. Sirtuin 1 expression will be evaluated since this has been reported to increase with resveratrol.
- 4. Other measurements: High performance liquid chromatography coupled with tandem mass spectrometry will be used to determine plasma and urine levels of resveratrol and its metabolites. In addition, urinary albumin/creatinine ratio, serum creatinine and estimated GFR will be assessed at the University of Iowa Clinical Lab.

# Statistical analysis

Normally distributed data are presented as mean±SD, non-normally distributed data as median (interquartile range), and categorical data as count (percentage of patients). To determine the effects of resveratrol supplementation on our primary and secondary outcomes, a generalized linear mixed effects model was used to examine the significance of condition, time, and their interaction for normally distributed variables, and a gamma mixed effects model was used for non-normally distributed variables. In each model, a random intercept was built for each patient to account for inherent between-patient variability. A complete case analysis was utilized when analyzing primary and secondary outcomes. A Wilcoxon Rank Sum Test was used to test differences in resveratrol metabolites between the resveratrol and placebo arms. Significance was set at an alpha level of 0.05. All analyses were performed in R, version 4.2.3 (R Foundation for Statistical Computing, Vienna, Austria).

#### References

- 1. Keith DS, Nichols GA, Gullion CM, Brown JB, and Smith DH. Longitudinal follow-up and outcomes among a population with chronic kidney disease in a large managed care organization. *Arch Intern Med.* 2004;164(6):659-63.
- 2. Brantsma AH, Bakker SJ, Hillege HL, de Zeeuw D, de Jong PE, and Gansevoort RT. Cardiovascular and renal outcome in subjects with K/DOQI stage 1-3 chronic kidney disease: the importance of urinary albumin excretion. *Nephrol Dial Transplant*. 2008;23(12):3851-8.
- 3. Go AS, Chertow GM, Fan D, McCulloch CE, and Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. *N Engl J Med.* 2004;351(13):1296-305.
- 4. McCullough PA, Jurkovitz CT, Pergola PE, McGill JB, Brown WW, Collins AJ, Chen SC, Li S, Singh A, Norris KC, et al. Independent components of chronic kidney disease as a cardiovascular risk state: results from the Kidney Early Evaluation Program (KEEP). *Arch Intern Med.* 2007;167(11):1122-9.
- 5. McCullough PA, Li S, Jurkovitz CT, Stevens L, Collins AJ, Chen SC, Norris KC, McFarlane S, Johnson B, Shlipak MG, et al. Chronic kidney disease, prevalence of premature cardiovascular disease, and relationship to short-term mortality. *Am Heart J.* 2008;156(2):277-83.
- 6. Weiner DE, Tighiouart H, Stark PC, Amin MG, MacLeod B, Griffith JL, Salem DN, Levey AS, and Sarnak MJ. Kidney disease as a risk factor for recurrent cardiovascular disease and mortality. *Am J Kidney Dis.* 2004;44(2):198-206.
- 7. Pálsson R, and Patel UD. Cardiovascular Complications of Diabetic Kidney Disease. *Advances in chronic kidney disease*. 2014;21(3):273-80.
- 8. Tuttle KR, Bakris GL, Bilous RW, Chiang JL, de Boer IH, Goldstein-Fuchs J, Hirsch IB, Kalantar-Zadeh K, Narva AS, Navaneethan SD, et al. Diabetic Kidney Disease: A Report From an ADA Consensus Conference. *Diabetes Care*. 2014;37(10):2864-83.
- 9. Csiszar A, Smith K, Labinskyy N, Orosz Z, Rivera A, and Ungvari Z. Resveratrol attenuates TNF-alpha-induced activation of coronary arterial endothelial cells: role of NF-kappaB inhibition. *Am J Physiol Heart Circ Physiol.* 2006;291(4):H1694-9.
- 10. Wallerath T, Deckert G, Ternes T, Anderson H, Li H, Witte K, and Forstermann U. Resveratrol, a polyphenolic phytoalexin present in red wine, enhances expression and activity of endothelial nitric oxide synthase. *Circulation*. 2002;106(13):1652-8.
- 11. Pellegatta F, Bertelli AA, Staels B, Duhem C, Fulgenzi A, and Ferrero ME. Different short- and long-term effects of resveratrol on nuclear factor-kappaB phosphorylation and nuclear appearance in human endothelial cells. *Am J Clin Nutr.* 2003;77(5):1220-8.
- 12. Sato M, Ray PS, Maulik G, Maulik N, Engelman RM, Bertelli AA, Bertelli A, and Das DK. Myocardial protection with red wine extract. *J Cardiovasc Pharmacol*. 2000;35(2):263-8.
- 13. Yousuf S, Atif F, Ahmad M, Hoda N, Ishrat T, Khan B, and Islam F. Resveratrol exerts its neuroprotective effect by modulating mitochondrial dysfunctions and associated cell death during cerebral ischemia. *Brain Res.* 2009;1250(242-53.
- 14. Faghihzadeh F, Adibi P, and Hekmatdoost A. The effects of resveratrol supplementation on cardiovascular risk factors in patients with non-alcoholic fatty liver disease: a randomised, double-blind, placebo-controlled study. *Br J Nutr.* 2015;114(5):796-803.

- 15. Thazhath SS, Wu T, Bound MJ, Checklin HL, Standfield S, Jones KL, Horowitz M, and Rayner CK. Administration of resveratrol for 5 wk has no effect on glucagon-like peptide 1 secretion, gastric emptying, or glycemic control in type 2 diabetes: a randomized controlled trial. *Am J Clin Nutr.* 2016;103(1):66-70.
- 16. Celermajer DS, Sorensen K, Ryalls M, Robinson J, Thomas O, Leonard JV, and Deanfield JE. Impaired endothelial function occurs in the systemic arteries of children with homozygous homocystinuria but not in their heterozygous parents. *J Am Coll Cardiol*. 1993;22(3):854-8.
- 17. Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, et al. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. *J Am Coll Cardiol*. 2002;39(2):257-65.
- 18. Jalal DI, Jablonski KL, McFann K, Chonchol MB, and Seals DR. Vascular endothelial function is not related to serum uric acid in healthy adults. *Am J Hypertens*. 2012;25(4):407-13.